CLINICAL TRIAL: NCT05457543
Title: Collection of Blood Products for Use in the Development and Validation of Point-of-Care In Vitro Diagnostic Liver Function Test Devices
Brief Title: Blood Collection for Development and Validation of Point-of-Care Diagnostic Liver Function Tests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Group K Diagnostics Inc. (Industry)
Responsible Party: Principal Investigator, Laura M Ferguson, PhD, Chief Scientific Officer, Group K Diagnostics Inc.
Other Study IDs: GKD001
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Liver Diseases; Healthy; Liver Cirrhosis; Liver Fibrosis
Keywords: liver function; diagnostic test; point of care
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood (not retained after testing), serum tested and retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult: A venous blood and capillary blood collection is taken from each participant and tested with investigative diagnostic tests.
  Interventions: Diagnostic Test: Adult

INTERVENTIONS:
Diagnostic Test: Adult — Investigational use of a novel liver function diagnostic test that involves a paper-based test device and a smartphone application.

SUMMARY:
This is an observational study exploring the performance of a novel point-of-care diagnostic testing platform designed to quantitate the presence of liver function biomarkers such as bilirubin. Blood samples will be collected from participants to further development and validation of the testing platform to support FDA review. The diagnostic device is intended to provide rapid in-office test results using a finger stick of blood, a reaction test device, and a smartphone app.

DETAILED DESCRIPTION:
The nature of outpatient diagnostics delays diagnosis and proper treatment due to the need to travel to a sample collection site that is designed for volume testing adding the individual's sample to the testing que. The physical and temporal separation of diagnostic testing from medical office or virtual care visits delays physician decision-making until results are available. Many patients even skip the recommended testing due to time and financial costs.

Many acute and chronic conditions result in disruption of normal liver function. Common prescription and over-the-counter medications also affect liver function when taken over extended periods or at elevated doses. Having multiple rapid, easy-to-use diagnostic tests on a single platform could improve condition diagnosis and medication monitoring by ensuring current test results are available every time and anywhere they could be useful for immediate medical decision-making.

This study will provide fresh blood samples for further development and validation of a novel point-of-care diagnostic testing platform. Tests for liver function biomarkers such as bilirubin, ALT (alanine transaminase), and AST (aspartate aminotransferase) will be characterized and validated using fresh whole blood, freshly prepared serum, and frozen serum. Enrolled participants will have a standard venous and a standard finger stick blood collection. Enrolled participants can return once weekly for blood draws or can chose to have only a single study visit. The study will continue until sufficient data has been generated to support review of the tests by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Able to read and understand an informed consent form written in English

Exclusion Criteria:

* Pregnancy
* Participated in the present study within the last 6 days
* Subject is subjectively unwell at the time of enrollment visit
* Subject previously participated and has asked to be withdrawn from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Regression analysis of bilirubin test results | 6 months
  Regression and other statistical analyses will be applied to bilirubin tests results to evaluate quantitation linearity, precision, and accuracy relative to a predicate device.

SECONDARY OUTCOMES:
Sensitivity of image analysis to changes in concentration of test analyte | 9 months
  Investigational device compositions will be evaluated for the resolution of colorimetric change as read by image analysis as the concentration of test analyte changes.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Ferguson, PhD, Principal Investigator — Group K Diagnostics Inc.
Locations (1):
- Group K Diagnostics, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AuYoung B, Gutha Ravichandran A, Patel D, Dave N, Shah A, Wronko-Stevens B, Bettencourt F, Rajan R, Menon N. A Low-Cost Paper-Based Device for the Colorimetric Quantification of Bilirubin in Serum Using Smartphone Technology. Front Chem. 2022 Jul 7;10:869086. doi: 10.3389/fchem.2022.869086. eCollection 2022. PMID 35873049

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT05457543/Prot_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT05457543/ICF_001.pdf